CLINICAL TRIAL: NCT01484548
Title: A Phase 1, Randomized Clinical Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of The LEISH-F3 + GLA-SE Vaccine Compared To The LEISH-F3 Protein Alone In Healthy Adult Subjects
Brief Title: Phase 1 LEISH-F3 Vaccine Trial in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IDRI-LVVPX-111
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine: 20 ug LEISH-F3 + 2 ug GLA-SE (Experimental): Low dose of adjuvant.
  Interventions: Biological: LEISH-F3 + GLA-SE
- Vaccine: 20 ug LEISH-F3 + 5 ug GLA-SE (Experimental): Higher dose of adjuvant.
  Interventions: Biological: LEISH-F3 + GLA-SE
- 20 ug LEISH-F3 alone (Active Comparator): 20 ug of LEISH-F3 antigen alone. 3 injections at Days 0, 28, and 56.
  Interventions: Biological: LEISH-F3 alone

INTERVENTIONS:
Biological: LEISH-F3 + GLA-SE — 20 ug of LEISH-F3 and 2 ug of GLA-SE adjuvant. 3 injections at Days 0, 28, and 56.
  Arms: Vaccine: 20 ug LEISH-F3 + 2 ug GLA-SE
Biological: LEISH-F3 + GLA-SE — 20 ug of LEISH-F3 and 5 ug of GLA-SE adjuvant. 3 injections at Days 0, 28, and 56.
  Arms: Vaccine: 20 ug LEISH-F3 + 5 ug GLA-SE
Biological: LEISH-F3 alone — 20 ug of LEISH-F3 antigen alone. 3 injections at Days 0, 28, and 56.
  Arms: 20 ug LEISH-F3 alone

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immunogenicity in healthy adult subjects of an investigational vaccine being developed for the prophylaxis of visceral leishmaniasis. The vaccine, identified as LEISH-F3 + GLA-SE, consists of the recombinant two-antigen Leishmania recombinant protein LEISH-F3 together with the adjuvant GLA-SE.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following criteria to be eligible for inclusion in the study:

* Males and females 18 years to 45 years of age.
* Must be in good general health as confirmed by a medical history and physical exam.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test on the day of each study injection, must not be breast-feeding, and are required to use one of the following methods of contraception during the first 3 months of the study: hormonal (e.g. oral, transdermal, intravaginal, implant, or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); abstinence; or bilateral tubal ligation (if no conception post-procedure). These precautions are necessary due to unknown effects that LEISH-F3 + GLA SE or LEISH-F3 alone might have in a fetus or newborn infant.
* The following screening laboratory blood tests must have values within the normal ranges or not clinically significant as determined by the PI and Medical Monitor: sodium, potassium, BUN, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, fasting glucose, fasting lipid panel, total WBC count, hemoglobin, and platelet count.
* The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
* Negative urine test for recreational drugs and alcohol per Clinical Research Unit standards.
* Urinalysis not clinically significant as determined by the study clinician.
* Must be capable of completing a study diary in English.
* Must give written informed consent, be able and willing to attend all evaluation visits, be reachable by telephone or personal contact by the study site personnel, and have a permanent address.

Exclusion Criteria:

Subjects who meet ANY of the following criteria will be excluded from the study (ineligible):

* History of possible infection with Leishmania or previous exposure to Leishmania vaccines or experimental products containing GLA-SE.
* Veterans who served in the military in the Middle East (Iran, Iraq), Afghanistan, or any other areas endemic to Leishmania.
* Travelers to, or immigrants from, areas endemic to Leishmania.
* Participation in another experimental protocol or receipt of any investigational products within the past 3 months.
* Treatment with immunosuppressive drugs (e.g., oral or injected steroids, such as prednisone; high dose inhaled steroids) or cytotoxic therapies (e.g., chemotherapy drugs or radiation) within the past 6 months.
* Received a blood transfusion within the past 3 months.
* Donated blood products (platelets, whole blood, plasma, etc.) within past 1 month.
* Received any vaccine within past 1 month. Note: No immunizations while on study with the exception of seasonal influenza vaccine which should not be given until 1 month after the third study injection (Day 84).
* History of autoimmune disease or other causes of immunosuppressive states.
* History or evidence of any acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic, or renal disorders, controlled hypertension), or use of medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Rash, tattoos or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
* BMI greater than 30 kg/m2
* Hypertension (systolic greater than 150 or diastolic greater than 95).
* History of significant psychiatric illness with current use of medication.
* Known or suspected alcohol or drug abuse within the past 6 months.
* Chronic smoker (less than 20 pack years).
* Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines, eggs, or unknown allergens.
* Subjects who are unlikely to cooperate with the requirements of the study protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events. | 421 days
  To evaluate the safety and tolerability of 20 μg of LEISH-F3 together with 2 or 5 μg of GLA-SE compared to 20 µg of LEISH-F3 alone following intramuscular administration on Days 0, 28, and 56. The safety assessments will be based on local and systemic reactions, including reported adverse events, changes in laboratory values, and changes in vital signs. The severity and relationship to treatment will be recorded for all adverse events.

SECONDARY OUTCOMES:
Immunogenicity | Days 0, 7, 35, 63, 84, and 168.
  To assess the immunogenicity of LEISH-F3 + GLA-SE compared to LEISH-F3 alone by evaluating IgG antibody and T-cell responses to LEISH-F3 at specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Piazza, MD, MPH, Study Director — Access to Advanced Health Institute (AAHI)
Locations (1):
- Comprehensive Clinical Development NW, Inc., Tacoma, Washington, United States